CLINICAL TRIAL: NCT02098772
Title: A Prospective Randomized Double Blind Multicenter Phase III Study Comparing Two Methods of Cardioplegia in Aortic Valve Surgery Custodiol-N Versus Custodiol
Brief Title: Phase III Study Comparing Two Methods of Cardioplegia in Aortic Valve Surgery Custodiol-N Versus Custodiol
Acronym: Custodiol-AV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. F. Köhler Chemie GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: CL-N-CSM-AV-III/05/12
Record Dates: First submitted 2014-02-14; First posted 2014-03-28 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2018-02

CONDITIONS: Aortic Valve Disease; Coronary Artery Disease (CAD)
Keywords: aortic valve disease; coronary bypass surgery; cardioplegic solutions
MeSH Terms: conditions — Aortic Valve Disease; Coronary Artery Disease | interventions — Custodiol-N solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Custodiol-N (Experimental): comparison of two cardioplegic solutions, Custodiol-N versus Custodiol, in aortic valve surgery
  Interventions: Drug: Custodiol-N
- Custodiol (Active Comparator): comparison of two cardioplegic solutions, Custodiol-N versus Custodiol, in aortic valve surgery
  Interventions: Drug: Custodiol

INTERVENTIONS:
Drug: Custodiol-N — comparison of two cardioplegic solutions, Custodiol-N versus Custodiol, in aortic valve surgery
  Arms: Custodiol-N
Drug: Custodiol — comparison of two cardioplegic solutions, Custodiol-N versus Custodiol, in aortic valve surgery
  Arms: Custodiol

SUMMARY:
The objective of this investigation is to compare the cardioprotective effects and safety of two cardioplegic solutions, HTK Cardioplegic Solution (Custodiol) and Custodiol-N in patients undergoing aortic valve surgery. The study design is a prospective, double blind, multicenter, randomized, Phase III comparison study intended to demonstrate superiority in surgical outcome between Custodiol and Custodiol-N as determined by CK-MB peak value 4-24 hours after opening of the aortic cross-clamp (primary endpoint), catecholamine requirement (cumulative dose) and cardiac Troponin T, occurrence of comorbid events postoperatively (e.g., myocardial infarction).

ELIGIBILITY:
Inclusion Criteria:

* Patients >/= 30 and </= 85 years of age
* Male or female with aortic valve disease
* Able to understand character and individual consequences of the clinical trial and to provide written informed consent to participate in the study
* Women of childbearing potential (ie, those who have not undergone a hysterectomy or who have not been post-menopausal for at least 12 consecutive months) must test negative for pregnancy prior to bypass surgery.

Exclusion Criteria:

* History of recent (< 6 weeks) Q-wave myocardial infarction
* Left ventricular ejection fraction < 25% (as assessed by any one of the following: contrast ventriculography, multigated acquisition scanning [MUGA], or 2-D ECHO)
* Patients on intra-aortic balloon devices or with history of previous coronary artery bypass surgery
* Pregnant or lactating patients
* Patients who have participated in any other investigational studies within 30 days previous to enrollment
* Patients in cardiogenic shock (defined as a systolic BP < 90 mmHg for over one hour despite inotropic and chronotropic support)
* Patients with severe chronic obstructive lung disease (FEV1 < 50%)
* Previous cardiac valvular disease (clinical relevant)
* GFR <60 ml/min
* Planned Ross-procedure, Mitral valve surgery, Aortic valve reconstruction, double valve surgery, other concomitant operations excluding coronary artery bypass surgery or closing a patent foramen ovale
* Evidence of severe organic (e.g. cirrhosis of the liver) or psychiatric disease by history or physical examination
* History of alcohol abuse, illicit drug use, significant mental illness, physical dependence to any opioid, or any history of drug abuse or addiction within 12 months of study enrollment.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2018-11-16 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
peak value for CK-MB | measured at 4, 8, 12, 16, 20 and 24 hours after the release of the aortic cross clamp

SECONDARY OUTCOMES:
Catecholamine requirement on SICU | within 24 hours (cumulative dose)

OTHER OUTCOMES:
Safety parameters | from time of the study inclusion up to the follow-up visit on day 5
  documentation and reporting of AE and SAE

CONTACTS AND LOCATIONS:
Overall Officials: Gabor Szabó, Prof., Principal Investigator — Department of Cardiac Surgery, University of Heidelberg, Im Neuenheimer Feld 110, 69120 Heidelberg
Locations (6):
- Germany (6):
  - Klinik für Herzchirurgie, Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Klinik für Herz- und Gefäßchirurgie GmbH, Herz-Kreislauf-Zentrum Rotenburg, Rotenburg an der Fulda, Hesse
  - Klinik für Herzchirurgie Universität Leipzig/ Herzzentrum Leipzig, Leipzig, Saxony
  - Klinik für Herz- und Thoraxchirurgie Universitätsklinikum Jena, Jena, Thuringia
  - Klinik für Thorax-, Herz- und Gefäßchirurgie, Uniklinik der RWTH Aachen, Aachen
  - Klinik für Gefäßchirurgie, Universitäres Herzzentrum am UKE Hamburg, Hamburg